CLINICAL TRIAL: NCT02616692
Title: Patient Preferences for Treatments for Hepatocellular Cancer (HCC) in Japan
Brief Title: HCC Patient Preferences in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18234
Record Dates: First submitted 2015-09-28; First posted 2015-11-30 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Cancer
Keywords: HCC; Patient preferences
MeSH Terms: conditions — Liver Neoplasms; Patient Preference | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCC patients / Cohort 1: Patient preferences associated with oral anti-cancer therapy (Sorafenib), repeated TACE, and HAIC and their perceptions regarding the respective treatment characteristics
  Interventions: Drug: Hepatocellular Cancer (HCC) treatments including oral anti-cancer therapy [Nexavar (Sorafenib, BAY43-9006)]

INTERVENTIONS:
Drug: Hepatocellular Cancer (HCC) treatments including oral anti-cancer therapy [Nexavar (Sorafenib, BAY43-9006)] — Oral anti-cancer therapy (Sorafenib, an multiple kinase inhibitor), repeated transarterial chemoembolization (TACE) procedures, and hepatic arterial infusion chemotherapy (HAIC)

SUMMARY:
This non-interventional cross-sectional online survey will evaluate preferences among patients with self-reported HCC. The survey will ask patients to express their preferences regarding descriptions of HCC treatments, which will include sorafenib (which will be described as 'oral anti-cancer therapy'), repeated transarterial chemoembolization (TACE), and hepatic arterial infusion chemotherapy (HAIC). Please note that all interventions that patients may have received before completing this online survey were given regardless of their participation in this survey. Questions also include asking patients to rank various treatment characteristics (e.g., mechanism of action, risk of adverse effects, etc.) relative to each other. The ultimate goal is to better understand patient perceptions of these treatments and to provide evidence to help in patients' and physicians' treatment decision-making in HCC.

ELIGIBILITY:
Inclusion Criteria:

The following eligibility criteria will be used:

* Have a diagnosis of HCC
* Are > 20 years of age
* Reside in Japan
* Are able to read and understand Japanese to provide informed consent and complete the survey instrument

Exclusion Criteria:

None are currently considered

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular cancer (HCC)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

PRIMARY OUTCOMES:
Preference weight scores for 13 selected HCC treatment attributes associated with Sorafenib, repeated TACE, and HAIC | up to 8 weeks
  Best-Worst Scaling scores for each attribute:
  1. Prevents formation of new blood vessels
  2. 2 tablets twice a day
  3. Risk of hand-foot skin reaction
  4. Risk of diarrhea
  5. Risk of stopping treatment because of side effects
  6. Artery branches in liver are plugged
  7. Several hour medical procedure under sedation with hospitalization
  8. Medical procedure repeated when needed
  9. Risk of liver damage
  10. Ongoing chemotherapy drugs to the liver
  11. Container and a catheter implanted in the body
  12. Risk of fever, abdominal pain, and nausea
  13. Risk of complications with catheter

SECONDARY OUTCOMES:
Response to the direct preference elicitation item asking which is most preferred: oral anti-cancer therapy (Sorafenib), repeated TACE, and HAIC | up to 8 weeks
Like/dislike ratings of each treatment attribute (Extent of patients like or dislike of different treatment attributes) | up to 8 weeks
  Specific scale responses: dislike a lot, dislike, neither like or dislike, like, like a lot
Willingness to try oral anti-cancer therapy (Sorafenib), TACE, and HAIC | up to 8 weeks
  Rated on a 0-100 scales
Maximum acceptable risk of hand-foot skin reaction willing to take for oral anti-cancer therapy (Sorafenib) therapy that will stop cancer from getting worse for a specified period of time | up to 8 weeks
  Mean percentage acceptable risk on a scale from 0% (will not accept any risk of hand-foot skin reaction) to 100% (will definitely accept a risk of hand-foot skin reaction)
Maximum acceptable risk of life-threatening side effect willing to take for oral anti-cancer therapy (Sorafenib) therapy that will stop cancer from getting worse for a specified period of time | up to 8 weeks
  Mean percentage acceptable risk on a scale from 0% (will not accept any risk of life-threatening side effect) to 100% (will definitely accept a risk of life-threatening side effect)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan